CLINICAL TRIAL: NCT05584592
Title: A Randomized Controlled Trial of Integrated Early Palliative Care for Advanced Gastric Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2020-0636
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Advanced Gastric Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intergrate early palliatuve care + Conventional chemotherapy (Experimental)
  Interventions: Other: Intergrate early palliatuve care + Conventional chemotherapy
- Conventional chemotherapy (Active Comparator)
  Interventions: Other: Conventional chemotherapy

INTERVENTIONS:
Other: Intergrate early palliatuve care + Conventional chemotherapy — Sixty patients with gastric and pancreatic cancer will be eligible, and 30 patients will be randomly assigned to the exercise therapy + high protein supplement group and 30 patients to the exercise therapy + placebo supplement group.
  Arms: Intergrate early palliatuve care + Conventional chemotherapy
Other: Conventional chemotherapy — patients to receive routine palliative care when they want it or when it is needed by health care providers. In other words, if a patient assigned to the control group desires palliative care, they can receive conventional palliative care.
  Arms: Conventional chemotherapy

SUMMARY:
Cancer patients and their families constantly face physical, psychosocial, economic, and existential problems, but palliative care to solve and prevent them is currently applied only at a late stage in Korean medical practice, which and has many limitations in solving practical difficulties. In order to solve the physical, mental, social, and spiritual health problems experienced by cancer patients in a situation where the cancer incidence rate is increasing every year, the timing and standard of providing palliative care in consideration of the current medical reality and the current status of chemotherapy There is an urgent need for research on a valid medical basis for a new Korean-style early palliative care program.

Early palliative care intervention study in patients with advanced cancer (Zimmermann et al, Lancet, 2014) and comparative study of early versus delayed palliative care intervention in patients with advanced cancer [Project ENABLE III] (Bakitas et al, JCO, 2015) The study started the intervention immediately after diagnosis of advanced or metastatic cancer. This is done earlier than traditional hospice palliative care, and provides professional services to not only proactively manage symptoms and improve quality of life, but also identify and implement the preferences, values, goals, and needs of patients and families. Although there are studies on the effect of early palliative care in multicenters for patients with locally advanced/metastatic gastric cancer, in the case of studies conducted at multicenters, there is no way to standardize the quality of palliative care at each research institute, so the intervention group is passive treatment. In many cases, it is difficult to obtain homogeneous results when the control group is cross-mixed with the intervention group. Thus, several factors are well-controlled and systematically Through this study, it is necessary to verify the effect of early palliative care in patients with gastric cancer, which occurs the most every year in Koreans.

About 170 patients with advanced gastric cancer who were histologically or cytologically diagnosed with gastric cancer at the participating institution are targeted. About 170 recruited patients will be randomly assigned to two groups, the intervention group and the control group.

DETAILED DESCRIPTION:
* Recruitment of research subjects: Outpatients and inpatients who meet the criteria for research are explained about the research and recruited, and written consent is obtained.
* Random assignment: The intervention group and the control group will be assigned 1:1, and whether the recruited patients are HER2-positive (positive vs negative), systemic activity (ECOG 0-1 vs 2), anticancer order [1st line vs 2nd] line (1st chemotherapy PFS of more than 6 months in case of 2nd line vs. PFS of primary chemotherapy less than 6 months in case of 2nd line) was randomized as a stratification factor.
* Intervention group (integrated early palliative care): While receiving standard chemotherapy, with the first meeting with the palliative care team within 4 weeks of randomization, and during the course of treatment regularly, once every 3 weeks (± 1 week) for 12 weeks Provides advance care planning, symptom control, and palliative care for other mental, social and spiritual problems. In the baseline survey, information about the Eul palliative care center is provided.
* Control group (standard chemotherapy group): Allows patients to receive conventional palliative care when they want or need it by medical staff. In other words, if a patient assigned to a control group desires palliative care, they can receive conventional palliative care.
* Data collection: The first questionnaire was conducted at the time of registration of the study subjects, the follow-up questionnaire was conducted at about 12 weeks, and survival was investigated after 1 year. The first questionnaire and follow-up questionnaire surveyed quality of life (EORTC QLQ-C30, EORTC QOL-ST022) and emotional disorder (HADS-D/A)

  ?Data Management: Keeping the completed subject questionnaire and recording the case record.
* Outcome indicators: The primary outcome indicators are evaluated as changes in the patient's comprehensive quality of life (Trial Outcome Index=EORTC QLQ-C30 + EORTC QOL-ST022) at the time of enrollment and 12 weeks of follow-up. , anticancer side effects, survival period, and changes in skeletal muscle mass index as secondary outcome indicators

ELIGIBILITY:
Inclusion Criteria:

1. Has a histologically or cytologically advanced gastric cancer patients
2. Those who are 19 years of age or older 3. Those who belong to ECOG performance status 0~2

4. Those who are planning to undergo 1st or 2nd palliative chemotherapy 5. Those who wish to participate in the research

Exclusion Criteria:

1. Those who are judged by the doctor to be unable to conduct this investigation due to medically poor health conditions (shortness of breath, etc.)
2. Those who have previously received palliative care or are receiving palliative care

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Changes in patient's comprehensive quality of life composite | 12 weeks
  Changes in patient's comprehensive quality of life (Trial Outcome Index=EORTC QLQ-C30 + EORTC QOL-ST022) at enrollment and 12-week follow-up The primary endpoint of this study was the change in the patient's comprehensive quality of life (Trial Outcome Index=EORTC QLQ-C30 + EORTC QOL-ST022) compared to the baseline outcome at week 12. The amount of change in the results at 12 weeks compared to the baseline result of the comprehensive quality of life (TOI) will be estimated in each group, and the effect size will be estimated for the difference in the amount of change between the two groups.

SECONDARY OUTCOMES:
Enotional disorders(HASA-D/A) | 2 years
  Both the intervention group and the control group are evaluated by Questionnaire evaluation tool (HADS-D/A) .
Objective Response Rate (ORR) | 2 years
  Objective response rate is defined as the number of patients with at least one confirmed visit response of CR or PR.
Progression-Free Survival (PFS) | 2 years
  To evaluate the treatment effect of Integrated Early Palliative Care group vs standard chemotherapy group on progression-free survival (PFS) rate.
Overall Survival (OS) | 2 years
  The time from the date of first dose and the date of death from any cause.
Skeletal muscle mass index (Skeletal muscle mass index, SMI) changes | 2 years
  Both the intervention group and the control group are evaluated by measuring skeletal muscle mass index (SMI) through Inbody®

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No